CLINICAL TRIAL: NCT00146640
Title: A New Timed-Release Tablet Formulation of Prednisone Compared to Standard Prednisone in Patients With Rheumatoid Arthritis- A Randomized, Multi-Centre, Double-Blind, Active Controlled Study With Open Extension on the New Drug Only
Brief Title: Prednisone Timed-Release Tablet (TRT) Study: Modified-Release (MR) Formulation of Prednisone Compared to Standard Immediate-Release (IR) Prednisone in Participants With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMR 62215-003
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Results first posted 2018-05-29 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Rheumatoid Arthritis
Keywords: active disease; morning stiffness of joints; nighttime application of prednisone; modified release prednisone
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- MR Prednisone (Experimental): Participants will receive MR prednisone at bed time and placebo matching to IR prednisone in the morning. Total duration of double blind treatment will be 12 weeks.
  Interventions: Drug: MR Prednisone; Drug: Placebo - IR Prednisone
- IR Prednisone (Active Comparator): Participants will receive IR prednisone in the morning and placebo matching to MR prednisone at bed time. Total duration of double blind treatment will be 12 weeks.
  Interventions: Drug: IR Prednisone; Drug: Placebo - MR Prednisone

INTERVENTIONS:
Drug: MR Prednisone — Participants will receive tablets containing MR prednisone (to achieve the appropriate dose of 3-10 milligrams [mg] prednisone per day) at bed time.
  Arms: MR Prednisone
Drug: IR Prednisone — Participants will receive tablets containing IR prednisone (to achieve the appropriate dose of 3-10 mg prednisone per day) in the morning.
  Arms: IR Prednisone
Drug: Placebo - MR Prednisone — Participants will receive placebo matching to MR prednisone tablet at bed time.
  Arms: IR Prednisone
Drug: Placebo - IR Prednisone — Participants will receive placebo matching to IR prednisone tablet in the morning.
  Arms: MR Prednisone

SUMMARY:
The objective of this study is to investigate if low doses of prednisone MR formulation, given at night and, with active drug release at 2 am, are more effective in controlling joint stiffness, and other disease symptoms of rheumatoid arthritis than standard IR prednisone given in the morning.

ELIGIBILITY:
Inclusion Criteria:

* Active disease (inflammatory signs, erythrocyte sedimentation rate [ESR], C-reactive protein [CRP])
* Stable condition
* Stable basic treatments
* Morning stiffness on previous treatment with standard prednisone (below or equal to 10 mg per day) greater than or equal to (>/=) 45 minutes

Exclusion Criteria:

* All contra-indications for glucocorticoids
* Pregnancy
* Concomitant treatment with biologics
* Intra-articular injections or synovectomy within the previous 4 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2004-08-31 (Actual); Primary Completion 2007-01-31 (Actual); Study Completion 2007-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (24):
- Germany (15):
  - Research Site, Aachen
  - Research Site, Bad Kreuznach
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Erlangen
  - Research Site, Frankfurt am Main
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Jena
  - Research Site, Leipzig
  - Research Site, München
  - Research Site, Ratingen
  - Research Site, Rostock
- Poland (9):
  - Research Site, Bialystok
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Sopot
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wroclaw

REFERENCES:
- [Result] Alten R, Doring G, Cutolo M, Gromnica-Ihle E, Witte S, Straub R, Buttgereit F. Hypothalamus-pituitary-adrenal axis function in patients with rheumatoid arthritis treated with nighttime-release prednisone. J Rheumatol. 2010 Oct;37(10):2025-31. doi: 10.3899/jrheum.100051. Epub 2010 Aug 3. PMID 20682671
- [Result] Buttgereit F, Doering G, Schaeffler A, Witte S, Sierakowski S, Gromnica-Ihle E, Jeka S, Krueger K, Szechinski J, Alten R. Efficacy of modified-release versus standard prednisone to reduce duration of morning stiffness of the joints in rheumatoid arthritis (CAPRA-1): a double-blind, randomised controlled trial. Lancet. 2008 Jan 19;371(9608):205-14. doi: 10.1016/S0140-6736(08)60132-4. PMID 18207016

RESULTS

PARTICIPANT FLOW:
Groups:
- MR Prednisone: Participants received tablets containing modified-release (MR) prednisone (to achieve the appropriate dose of 3-10 milligrams [mg] prednisone per day) at bed time and placebo matching to immediate-release (IR) prednisone tablet in the morning. Total duration of double blind treatment was 12 weeks.
- IR Prednisone: Participants received tablets containing IR prednisone (to achieve the appropriate dose of 3-10 mg prednisone per day) in the morning and placebo matching to MR prednisone tablet at bed time. Total duration of double blind treatment was 12 weeks.
Period: Overall Study
Arm/Group | MR Prednisone | IR Prednisone
Started | 144 | 144
Completed | 121 | 130
Not Completed | 23 | 14
Not completed — Adverse Event | 12 | 10
Not completed — Medical Reasons | 3 | 0
Not completed — Non-Medical Reasons | 8 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all randomized participants.
Groups:
- MR Prednisone: Participants received tablets containing MR prednisone (to achieve the appropriate dose of 3-10 mg prednisone per day) at bed time and placebo matching to IR prednisone tablet in the morning. Total duration of double blind treatment was 12 weeks.
- Total: Total of all reporting groups
Arm/Group | MR Prednisone | IR Prednisone | Total
Number analyzed (Participants) | 144 | 144 | 288
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (11.2) | 55.4 (11.4) | 55.0 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 122 | 247
  Male | 19 | 22 | 41

OUTCOME MEASURES:

1. Primary Outcome: Relative Change From Baseline in Duration of Morning Stiffness at Week 12
Description: Duration of morning stiffness was defined as the time elapsed (in minutes) between the time of usual awakening (even if not in the morning) and the time the participant was able to resume normal activities without stiffness. Relative (percent) change = ([value at Week 12 minus value at Baseline] divided by [value at baseline]) multiplied by 100.
Time Frame: Baseline, Week 12
Population: ITT Population. Here, overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | MR Prednisone | IR Prednisone
Number analyzed (Participants) | 125 | 129
percent change | -22.7 (89.1) | -0.4 (89.0)

2. Secondary Outcome: Relative Change From Baseline in 28-Joint Disease Activity Score (DAS28) at Week 12
Description: DAS28 calculated from the number of swollen joints (SJC) and painful joints (PJC) using the 28 joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and patient's global assessment (PGA) of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). Total DAS28 score range from 0 to approximately 10. DAS28 less than or equal to (≤) 3.2 = low disease activity, DAS28 greater than (>) 3.2 to 5.1 = moderate to high disease activity, and DAS28 >5.1 = severe disease activity. Relative (percent) change = ([value at Week 12 minus value at Baseline] divided by [value at baseline]) multiplied by 100.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | MR Prednisone | IR Prednisone
Number analyzed (Participants) | 136 | 137
percent change | -9.03 [-11.9 to -6.2] | -12.30 [-15.2 to -9.4]

3. Secondary Outcome: Percentage of Participants With Recurrence of Joint Stiffness at Week 12
Description: Participants recorded the status of recurrence of joint stiffness (Yes/No) in diary data. Percentage of participants who selected Yes for recurrence of joint stiffness, are reported.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | MR Prednisone | IR Prednisone
Number analyzed (Participants) | 119 | 127
percentage of participants | 47 | 43

4. Secondary Outcome: Relative Change From Baseline in Pain Intensity at Week 12
Description: Participants assessed pain intensity on a 100 millimeter (mm) visual analog scale (VAS), where 0 mm = no pain, 100 mm = worst pain. Relative (percent) change = ([value at Week 12 minus value at Baseline] divided by [value at baseline]) multiplied by 100.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | MR Prednisone | IR Prednisone
Number analyzed (Participants) | 141 | 143
percent change | -8.57 [-17.7 to 0.6] | -6.53 [-20.4 to 7.3]

5. Secondary Outcome: Relative Change From Baseline in Quality of Sleep at Week 12
Description: Participants assessed quality of sleep on a 100 mm VAS, where 0 mm = very good, 100 mm = very bad. Relative (percent) change = ([value at Week 12 minus value at Baseline] divided by [value at baseline]) multiplied by 100.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | MR Prednisone | IR Prednisone
Number analyzed (Participants) | 141 | 143
percent change | 4.63 [-9.9 to 19.1] | 0.13 [-12.3 to 12.5]

6. Secondary Outcome: Relative Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 12
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty. Relative (percent) change = ([value at Week 12 minus value at Baseline] divided by [value at baseline]) multiplied by 100.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | MR Prednisone | IR Prednisone
Number analyzed (Participants) | 137 | 138
percent change | 0.07 [-6.6 to 6.7] | -4.7 [-9.6 to 0.1]

7. Secondary Outcome: Relative Change From Baseline in Short-Form 36 (SF36) Mental Component Score (MCS) at Week 12
Description: SF-36 is a standardized survey evaluating 8 domains of functional health and wellbeing: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a domain was an average of the individual question scores, which were scaled 0-100 (100=highest level of functioning). Score from mental health, role emotional, social functioning, and vitality domains were averaged to calculate MCS. Total score range for MCS was 0-100 (100=highest level of mental functioning). Relative (percent) change = ([value at Week 12 minus value at Baseline] divided by [value at baseline]) multiplied by 100.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | MR Prednisone | IR Prednisone
Number analyzed (Participants) | 114 | 117
percent change | 10.63 [0.8 to 20.5] | 18.08 [9.7 to 26.4]

8. Secondary Outcome: Relative Change From Baseline in SF36 Physical Component Score (PCS) at Week 12
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and wellbeing: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a domain was an average of the individual question scores, which were scaled 0-100 (100=highest level of functioning). Score from physical function, role physical, bodily pain, and general health domains were averaged to calculate PCS. Total score range for PCS was 0-100 (100=highest level of physical functioning). Relative (percent) change = ([value at Week 12 minus value at Baseline] divided by [value at baseline]) multiplied by 100.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | MR Prednisone | IR Prednisone
Number analyzed (Participants) | 114 | 117
percent change | 19.43 [7.77 to 31.1] | 21.0 [11.05 to 30.9]

ADVERSE EVENTS:
Description: Among serious adverse events (SAEs), only data for total # affected by any SAE is available. Due diligence was done and all potential information sources have been exhausted; no further information could be retrieved. Hence, for SAEs the preferred term is reported as "Not Available" and System Organ Class as "General Disorders".
Arm/Group | MR Prednisone | IR Prednisone
Serious Adverse Events (participants affected / at risk) | 4/144 | 3/144
Other Adverse Events (participants affected / at risk) | 20/144 | 29/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MR Prednisone (N=144) | IR Prednisone (N=144)
(General disorders) | 4 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MR Prednisone (N=144) | IR Prednisone (N=144)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Rheumatoid arthritis (Immune system disorders) | 11 | 13
Abdominal pain (upper) (Gastrointestinal disorders) | 5 | 8

LIMITATIONS AND CAVEATS:
For SAEs, due diligence was done and all potential information sources have been exhausted, no further information could be retrieved apart from what is currently reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No